CLINICAL TRIAL: NCT01521884
Title: Longitudinal Changes In Fatigue And Health Status (aims2) In Ra Patients Treated With Sc Anti-tnf-alpha Therapy
Brief Title: Study Looking at Longitudinal Changes in Fatigue and Health Status in Rheumatoid Arthritis (RA) Patients Treated With Subcutaneous Anti-TNF-α Therapy
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0881A1-4748; B1801046 (Other: Alias Study Number)
Record Dates: First submitted 2011-08-19; First posted 2012-01-31 (Estimated); Results first posted 2015-02-19 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2015-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- RA Patients treated with SC anti-TNF
  Interventions: Other: SC anti-TNF

INTERVENTIONS:
Other: SC anti-TNF — SC anti-TNF

SUMMARY:
People affected by rheumatoid arthritis are often suffering from fatigue and decreased QOL. In this study we are measuring the impact of SC biologics on these parameters.

DETAILED DESCRIPTION:
Observational prospective study Purely descriptive

ELIGIBILITY:
Inclusion Criteria:

Patients who:

* Are active RA patients (as judged by treating MD)
* Are 18 years of age or older at time of consent
* Are scheduled by their rheumatologist to initiate SC anti-TNF-α therapy + MTX

Exclusion Criteria:

Use of biologics (or any experimental drug) in the last 3 months before initiation of SC anti-TNF-α therapy.

Participation in other clinical or observational trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients seen in a rheumatology practice
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2010-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- UZ Gasthuisberg, Leuven, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0881A1-4748&StudyName=Study%20Looking%20at%20Longitudinal%20Changes%20in%20Fatigue%20and%20Health%20Status%20in%20Rheumatoid%20Arthritis%20%28RA%29%20Patients%20Treated%20with%20Subcutaneous%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Anti-Tumour Necrosis Factor Alpha (Anti-TNF-alpha): Participants with rheumatoid arthritis (RA), who received subcutaneous anti-TNF-alpha therapy along with methotrexate as per treating physician's discretion based on summary of product characteristics, were followed up for 2 years.
Period: Overall Study
Arm/Group | Anti-Tumour Necrosis Factor Alpha (Anti-TNF-alpha)
Started | 62
Completed | 35
Not Completed | 27
Not completed — Non Responders | 10
Not completed — Adverse Event | 5
Not completed — Pregnancy | 1
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 2
Not completed — Protocol Violation | 3
Not completed — Participant non-eligible | 1
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Population: Intention to treat (ITT) population included all participants for whom the primary endpoint or one of the secondary endpoints could be determined at baseline. Here "N" (Overall Number of Baseline Participants) includes participants with non-missing baseline data.
Arm/Group | Anti-Tumour Necrosis Factor Alpha (Anti-TNF-alpha)
Number analyzed (Participants) | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (11.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 15

OUTCOME MEASURES:

1. Primary Outcome: Arthritis Impact Measurement Scale - Version 2 (AIMS2) Main Component Score at Baseline
Description: AIMS2 is a disease-specific measure of physical, social, and emotional well-being. It is a 78-item questionnaire assessing 12 scales: moving capacities, walking and dexterity, hand and fingers movements, arm movements, self-care, household activities, social activities, support of family and friends, joint pain, work, nervous tension and psychological condition (anxiety and depression). Each item was scored as 0 (or 1, best situation) to 4 (worst situation). Sub-total score of each of the 12 scales normalized to a maximum of 10. Total score were calculated for AIMS2 Affect ([Level of tension + Mood]/2), AIMS2 Physical ([Mobility level + Walking and bending + Hand and finger function + Arm function + Self Care + Household tasks]/6), and AIMS2 Symptom (Arthritis pain) with total score range from 0 to 10 for all component scores, where higher scores indicated worse situation.
Time Frame: Baseline
Population: ITT population included participants for whom the primary endpoint or 1 of the secondary endpoints could be determined at baseline. Here "n" = participants who were evaluable for this measure for specified component score. The results for social interaction and role components of AIMS2 were not analyzed due to change in planned analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anti-Tumour Necrosis Factor Alpha (Anti-TNF-alpha)
Number analyzed (Participants) | 62
units on a scale
  AIMS2-Physical Score (n=59) | 3.5 (1.7)
  AIMS2-Affect Score (n=59) | 4.8 (1.7)
  AIMS2-Symptom Score (n=58) | 7.3 (1.8)

2. Primary Outcome: Arthritis Impact Measurement Scale - Version 2 (AIMS2) Main Component Score at Month 6
Description: as for outcome 1
Time Frame: Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anti-Tumour Necrosis Factor Alpha (Anti-TNF-alpha)
Number analyzed (Participants) | 62
units on a scale
  AIMS2-Physical Score (n=47) | 2.3 (1.7)
  AIMS2-Affect Score (n=49) | 3.8 (1.9)
  AIMS2-Symptom Score (n=49) | 5.1 (2.5)

3. Primary Outcome: Arthritis Impact Measurement Scale - Version 2 (AIMS2) Main Component Score at Month 12
Description: as for outcome 1
Time Frame: Month 12
Population: ITT population included participants for whom the primary endpoint or 1 of the secondary endpoints could be determined at baseline. Here "N" (number of participants analyzed) = participants who were evaluable for this measure. The results for social interaction and role components of AIMS2 were not analyzed due to change in planned analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anti-Tumour Necrosis Factor Alpha (Anti-TNF-alpha)
Number analyzed (Participants) | 42
units on a scale
  AIMS2-Physical Score | 2.1 (1.3)
  AIMS2-Affect Score | 3.5 (1.8)
  AIMS2-Symptom Score | 4.3 (2.7)

4. Primary Outcome: Arthritis Impact Measurement Scale - Version 2 (AIMS2) Main Component Score at Month 18
Description: as for outcome 1
Time Frame: Month 18
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anti-Tumour Necrosis Factor Alpha (Anti-TNF-alpha)
Number analyzed (Participants) | 62
units on a scale
  AIMS2-Physical Score (n=30) | 2.6 (1.7)
  AIMS2-Affect Score (n=31) | 3.4 (1.8)
  AIMS2-Symptom Score (n=31) | 4.5 (2.1)

5. Primary Outcome: Arthritis Impact Measurement Scale - Version 2 (AIMS2) Main Component Score at Month 24
Description: as for outcome 1
Time Frame: Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anti-Tumour Necrosis Factor Alpha (Anti-TNF-alpha)
Number analyzed (Participants) | 62
units on a scale
  AIMS2-Physical Score (n=31) | 2.2 (1.7)
  AIMS2-Affect Score (n=31) | 3.2 (1.9)
  AIMS2-Symptom Score (n=30) | 3.8 (2.3)

6. Secondary Outcome: Visual Analog Scale (VAS) Fatigue Score
Description: Participants recorded their fatigue score on a range of 0 to 10, where higher score indicated higher intensity of fatigue.
Time Frame: Baseline, Month 6, 12, 18, 24
Population: ITT population included participants for whom the primary endpoint or 1 of the secondary endpoints could be determined at baseline. Here "n" = participants who were evaluable for this measure for specified component score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anti-Tumour Necrosis Factor Alpha (Anti-TNF-alpha)
Number analyzed (Participants) | 62
units on a scale
  Baseline (n=56) | 6.4 (1.93)
  Month 6 (n=47) | 4.7 (2.43)
  Month 12 (n=42) | 4.4 (2.41)
  Month 18 (n=31) | 4.3 (2.04)
  Month 24 (n=30) | 4.6 (2.43)

7. Secondary Outcome: Disease Activity Score Based on 28-Joints Count and Erythrocyte Sedimentation Rate (DAS 28-ESR)
Description: DAS28-ESR was calculated from the number of swollen joints (SJC) and tender joints (TJC ) using the 28 joints count, the erythrocyte sedimentation rate (ESR) (millimeter per hour [mm/hour]) and participant's assessment of disease activity visual analog scale (scores ranging 0 [very well] to 100 mm [extremely bad]). Total score range: 0-10, higher score=more disease activity (DA). DAS28-ESR less than equal to (<=) 3.2 = low disease activity, DAS28 greater than (>) 3.2 to 5.1 = moderate to high DA
Time Frame: Baseline, Month 6, 12, 18, 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anti-Tumour Necrosis Factor Alpha (Anti-TNF-alpha)
Number analyzed (Participants) | 62
units on a scale
  Baseline (n=55) | 4.93 (1.27)
  Month 6 (n=41) | 3.21 (1.37)
  Month 12 (n=37) | 3.05 (1.28)
  Month 18 (n=24) | 3.04 (1.27)
  Month 24 (n=23) | 2.44 (1.11)

8. Secondary Outcome: Disease Activity Score Based on 28-Joints Count and C-Reactive Protein (DAS 28-CRP)
Description: DAS28-CRP was calculated from the number of swollen joints ( SJC) and tender joints (TJC) count using 28 joint count and CRP (milligram per liter [mg/L]). Total score range: 0-10, higher score= more disease activity. DAS28 (CRP) : <3.2= low disease activity, >3.2 to 5.1 = moderate to high disease activity and less than (<)2.6 = remission.
Time Frame: Baseline, Month 6, 12, 18, 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anti-Tumour Necrosis Factor Alpha (Anti-TNF-alpha)
Number analyzed (Participants) | 62
units on a scale
  Baseline (n=23) | 4.59 (1.28)
  Month 6 (n=21) | 2.50 (1.06)
  Month 12 (n=20) | 2.75 (1.27)
  Month 18 (n=21) | 2.59 (0.83)
  Month 24 (n=19) | 2.35 (1.11)

9. Secondary Outcome: Health Assessment Questionnaire (HAQ) Total Score
Description: HAQ: 20-item participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom, arise, eat, walk, reach, grip, hygiene and common activities. Each item scored on 4-point scale, 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as sum of item scores. HAQ total score was 0 to 60 (as used in Belgium), where greater score indicated greater difficulty.
Time Frame: Baseline, Month 6, 12, 18, 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anti-Tumour Necrosis Factor Alpha (Anti-TNF-alpha)
Number analyzed (Participants) | 59
units on a scale
  Baseline (n=59) | 30.17 (8.765)
  Month 6 (n=49) | 22.99 (7.524)
  Month 12 (n=44) | 22.45 (8.729)
  Month 18 (n=32) | 23.60 (6.794)
  Month 24 (n=31) | 22.84 (6.769)

10. Other Pre Specified Outcome: Spearman Correlation Coefficient Between Arthritis Impact Measurement Scale - Version 2 (AIMS2) Main Components and Visual Analog Scale (VAS) Fatigue Score
Description: Spearman correlation coefficient between AIMS2 component score and VAS fatigue score (AIMS2 component score versus [vs] VAS fatigue) was calculated. AIMS2 : 78-item questionnaire assessing 12 scales. Each item was scored as 0 (or 1, best situation) to 4 (worst situation). Sub-total score of each of the 12 scales normalized to a maximum of 10. Total score were calculated for AIMS2 Affect ([Level of tension + Mood]/2), AIMS2 Physical ([Mobility level + Walking and bending + Hand and finger function + Arm function + Self Care + Household tasks]/6), and AIMS2 Symptom (Arthritis pain); total score range from 0 to 10, higher scores indicates worse situation and VAS score: Participants recorded their fatigue score on a range of 0 to 10, where higher score indicated higher intensity of fatigue.
Time Frame: Baseline, Month 6, 12, 18, 24
Population: as for outcome 1
Measure: Number; unit: correlation coefficient
Arm/Group | Anti-Tumour Necrosis Factor Alpha (Anti-TNF-alpha)
Number analyzed (Participants) | 62
correlation coefficient
  Baseline: AIMS2 Physical vs VAS fatigue (n=56) | 0.497
  Baseline: AIMS2 Affect vs VAS fatigue (n=56) | 0.419
  Baseline: AIMS2 Symptom vs VAS fatigue (n=55) | 0.516
  Month 6: AIMS2 Physical vs VAS fatigue (n=45) | 0.617
  Month 6: AIMS2 Affect at vs VAS fatigue (n=47) | 0.714
  Month 6: AIMS2 Symptom vs VAS fatigue (n=47) | 0.624
  Month 12: AIMS2 Physical vs VAS fatigue (n=41) | 0.361
  Month 12: AIMS2 Affect vs VAS fatigue (n=41) | 0.365
  Month 12: AIMS2 Symptom vs VAS fatigue (n=41) | 0.330
  Month 18: AIMS2 Physical vs VAS fatigue (n=30) | 0.318
  Month 18: AIMS2 Affect vs VAS fatigue (n=31) | 0.428
  Month 18: AIMS2 Symptom vs VAS fatigue (n=31) | 0.376
  Month 24: AIMS2 Physical vs VAS fatigue (n=30) | 0.452
  Month 24: AIMS2 Affect vs VAS fatigue (n=30) | 0.591
  Month 24: AIMS2 Symptom vs VAS fatigue (n=29) | 0.429

11. Other Pre Specified Outcome: Pearson Correlation Coefficient Between Arthritis Impact Measurement Scale - Version 2 (AIMS2) Main Components and Disease Activity Score Based on 28-Joints Count and Erythrocyte Sedimentation (DAS 28-ESR)
Description: Pearson correlation coefficient between AIMS2 component score and DAS28-ESR score (AIMS2 component score vs DAS28-ESR) was calculated. AIMS2: 78-item questionnaire assessing 12 scales. Each item was scored as 0 (or 1, best situation) to 4 (worst situation). Sub-total score of each of the 12 scales normalized to a maximum of 10. Total score were calculated for AIMS2 Affect ([Level of tension + Mood]/2), AIMS2 Physical ([Mobility level + Walking and bending + Hand and finger function + Arm function + Self Care + Household tasks]/6), and AIMS2 Symptom (Arthritis pain); total score range from 0 to 10, higher scores indicates worse situation and DAS28-ESR calculated from the number of SJC and TJC using the 28 joints count, ESR (mm/hour) and participant's assessment of disease activity VAS (scores ranging 0 [very well] to 100 mm [extremely bad]). Total score range: 0-10, higher score= more disease activity. DAS28-ESR <= 3.2 = low DA, DAS28 > 3.2 to 5.1 = moderate to high DA.
Time Frame: Baseline, Month 6,1 2, 18, 24
Population: ITT population, Here "n" = participants evaluable for this measure for specified component score and "N" (number of participants analyzed) = participants who were evaluable for this measure. The results for social interaction and role components of AIMS2 were not analyzed due to change in planned analysis.
Measure: Number; unit: correlation coefficient
Arm/Group | Anti-Tumour Necrosis Factor Alpha (Anti-TNF-alpha)
Number analyzed (Participants) | 62
correlation coefficient
  Baseline: AIMS2 Physical vs DAS28-ESR (n=53) | 0.366
  Baseline: AIMS2 Affect vs DAS28-ESR (n=53) | 0.071
  Baseline: AIMS2 Symptom vs DAS28-ESR (n=52) | 0.427
  Month 6: AIMS2 Physical vs DAS28-ESR (n=38) | 0.254
  Month 6: AIMS2 Affect vs DAS28-ESR (n=40) | 0.561
  Month 6: AIMS2 Symptom vs DAS28-ESR (n=40) | 0.602
  Month 12: AIMS2 Physical vs DAS28-ESR (n=33) | 0.399
  Month 12: AIMS2 Affect vs DAS28-ESR (n=33) | 0.263
  Month 12: AIMS2 Symptom vs DAS28-ESR (n=33) | 0.285
  Month 18: AIMS2 Physical vs DAS28-ESR (n=20) | 0.334
  Month 18: AIMS2 Affect vs DAS28-ESR (n=21) | 0.205
  Month 18: AIMS2 Symptom vs DAS28-ESR (n=21) | 0.336
  Month 24: AIMS2 Physical vs DAS28-ESR (n=21) | 0.110
  Month 24: AIMS2 Affect vs DAS28-ESR (n=21) | 0.180
  Month 24: AIMS2 Symptom vs DAS28-ESR (n=20) | 0.233

12. Other Pre Specified Outcome: Pearson Correlation Coefficient Between Arthritis Impact Measurement Scale- Version 2 (AIMS2) Main Components and Disease Activity Score Based on 28-Joints Count and C-Reactive Protein (DAS 28-CRP)
Description: Pearson correlation coefficient between AIMS2 component score and DAS28-CRP score (AIMS2 component score vs DAS28-CRP) was calculated. AIMS2: 78-item questionnaire assessing 12 scales. Each item was scored as 0 (or 1, best situation) to 4 (worst situation). Sub-total score of each of the 12 scales normalized to a maximum of 10. Total score were calculated for AIMS2 Affect ([Level of tension + Mood]/2), AIMS2 Physical ([Mobility level + Walking and bending + Hand and finger function + Arm function + Self Care + Household tasks]/6), and AIMS2 Symptom (Arthritis pain); total score range from 0 to 10, higher scores indicates worse situation DAS28-CRP was calculated from the number of SJC and TJC count using 28 joint count and CRP (mg/L). Total score range: 0-10, higher score= more disease activity. DAS28 (CRP): <3.2= low DA, >3.2 to 5.1 = moderate to high DA and <2.6 = remission.
Time Frame: Baseline, Month 6, 12, 18, 24
Population: as for outcome 1
Measure: Number; unit: correlation coefficient
Arm/Group | Anti-Tumour Necrosis Factor Alpha (Anti-TNF-alpha)
Number analyzed (Participants) | 62
correlation coefficient
  Baseline: AIMS2 Physical vs DAS 28-CRP (n=22) | 0.014
  Baseline: AIMS2 Affect vs DAS 28-CRP (n=22) | 0.238
  Baseline: AIMS2 Symptom vs DAS 28-CRP (n=22) | 0.097
  Month 6: AIMS2 Physical vs DAS 28-CRP (n=19) | 0.443
  Month 6: AIMS2 Affect vs DAS 28-CRP (n=20) | 0.344
  Month 6: AIMS2 Symptom vs DAS 28-CRP (n=20) | 0.583
  Month 12: AIMS2 Physical vs DAS 28-CRP (n=19) | 0.697
  Month 12: AIMS2 Affect vs DAS 28-CRP (n=19) | 0.425
  Month 12: AIMS2 Symptom vs DAS 28-CRP (n=19) | 0.541
  Month 18: AIMS2 Physical vs DAS 28-CRP (n=16) | 0.554
  Month 18: AIMS2 Affect vs DAS 28-CRP (n=16) | 0.368
  Month 18: AIMS2 Symptom vs DAS 28-CRP (n=16) | 0.617
  Month 24: AIMS2 Physical vs DAS 28-CRP (n=18) | 0.494
  Month 24: AIMS2 Affect vs DAS 28-CRP (n=18) | 0.487
  Month 24: AIMS2 Symptom vs DAS 28-CRP (n=18) | 0.478

13. Other Pre Specified Outcome: Spearman Correlation Coefficient Between Disease Activity Score Based on 28-Joints Count and Erythrocyte Sedimentation (DAS 28-ESR) and Visual Analog Scale (VAS) Fatigue Score
Description: Spearman correlation coefficient between DAS28-ESR and VAS fatigue (DAS28-ESR vs VAS score) was calculated. DAS28-ESR calculated from the number of SJC and TJC using the 28 joints count, ESR (mm/hour) and participant's assessment of disease activity VAS (scores ranging 0 [very well] to 100 mm [extremely bad]). Total score range: 0-10, higher score= more disease activity. DAS28-ESR <= 3.2 = low DA, DAS28 > 3.2 to 5.1 = moderate to high DA and VAS fatigue = Participants recorded their fatigue score on a range of 0 to 10, where higher score indicated higher intensity of fatigue.
Time Frame: Baseline, Month 6, 12, 18, 24
Population: as for outcome 6
Measure: Number; unit: correlation coefficient
Arm/Group | Anti-Tumour Necrosis Factor Alpha (Anti-TNF-alpha)
Number analyzed (Participants) | 62
correlation coefficient
  Baseline: DAS28-ESR vs VAS fatigue (n=50) | 0.370
  Month 6: DAS28-ESR vs VAS fatigue (n=38) | 0.394
  Month 12: DAS28-ESR vs VAS fatigue (n=34) | 0.215
  Month 18: DAS28-ESR vs VAS fatigue (n=21) | 0.073
  Month 24: DAS28-ESR vs VAS fatigue (n=21) | 0.401

14. Other Pre Specified Outcome: Spearman Correlation Coefficient Between Disease Activity Score Based on 28-Joints Count and C-Reactive Protein (DAS 28-CRP) and Visual Analog Scale (VAS) Fatigue Score
Description: Spearman correlation coefficient between DAS28-CRP and VAS score (DAS28-CRP vs VAS score) was calculated. DAS28-CRP was calculated from the number of SJC and TJC count using 28 joint count and CRP (mg/L). Total score range: 0-10, higher score= more disease activity. DAS28 (CRP): <3.2= low DA, >3.2 to 5.1 = moderate to high DA and <2.6 = remission and VAS= Participants recorded their fatigue score on a range of 0 to 10, where higher score indicated higher intensity of fatigue.
Time Frame: Baseline, Month 6, 12, 18, 24
Population: as for outcome 6
Measure: Number; unit: correlation coefficient
Arm/Group | Anti-Tumour Necrosis Factor Alpha (Anti-TNF-alpha)
Number analyzed (Participants) | 62
correlation coefficient
  Baseline: DAS28-CRP vs VAS fatigue (n=22) | 0.096
  Month 6: DAS28-CRP vs VAS fatigue (n=19) | 0.291
  Month 12: DAS28-CRP vs VAS fatigue (n=19) | 0.271
  Month 18: DAS28-CRP vs VAS fatigue (n=16) | 0.193
  Month 24: DAS28-CRP vs VAS fatigue (n=17) | 0.300

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one subject and as non-serious in another subject, or one subject may have experienced both a serious and non-serious event during the study.
Arm/Group | Anti-Tumour Necrosis Factor Alpha (Anti-TNF-alpha)
Serious Adverse Events (participants affected / at risk) | 1/62
Other Adverse Events (participants affected / at risk) | 4/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anti-Tumour Necrosis Factor Alpha (Anti-TNF-alpha) (N=62)
Spondylodiscitis (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anti-Tumour Necrosis Factor Alpha (Anti-TNF-alpha) (N=62)
Asthma (General disorders) | 1
Tachycardia (General disorders) | 1
Headache (General disorders) | 1
Nausea (General disorders) | 1
Purulent rhinorrhea (General disorders) | 1

LIMITATIONS AND CAVEATS:
Designation of primary and secondary endpoints was based on study team's inputs, as the endpoints were not prioritized in the study protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.